CLINICAL TRIAL: NCT03473444
Title: Prevalence of Hyperuricemia in Pakistan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: OBS Pakistan (Industry)
Responsible Party: Sponsor
Other Study IDs: ZeroGout-OBS-002
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Hyperuricemia
Keywords: uric acid; prevalence; pakistan
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of hyperuricemia has rarely been investigated in developing countries Hyperuricemia, or raised serum uric acid (SUA), is the condition closely associated with gout due to the deposition of monosodium urate crystals in peripheral joints and soft tissues. Hyperuricemia is associated with an increased risk for incident hypertension, independent of traditional hypertension risk factors. This risk appears more pronounced in younger individuals and women. Cross-sectional studies show an association of hyperuricemia with the presence of CKD. Insulin resistance plays a potentially key role in the causal relationship between metabolic syndrome, type 2 Diabetes and hyperuricemia. Furthermore, it is likely that hyperuricemia and insulin resistance share a bidirectional causal effect. The rationale of this study is to determine prevalence of hyperuricemia in Pakistan.

DETAILED DESCRIPTION:
Informed consent will be obtained from all patients and their attendant coming to clinics. Those who will agree to be part of this study were asked a questionnaire about co-morbidity and symptoms.

Uric acid levels will be assessed by using UASure Blood Uric Acid Monitoring System. Male with uric acid levels greater than 7 mg/dl and female greater than 6 mg/dl were classified as hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent given

Exclusion Criteria:

* No Informed consent provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Informed consent was obtained from all patients and their attendant coming to clinics. Those who agreed to be part of this study were asked a questionnaire about co-morbidity and symptoms.
  Uric acid levels were assessed by using UASure Blood Uric Acid Monitoring System. Male with uric acid levels greater than 7 mg/dl and female greater than 6 mg/dl were classified as hyperuricemia.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Hyperuricemia | 4 weeks
  To find out the frequency uric acid levels in Pakistani general population

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abid Naeem, Mirpur, Azad Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No